CLINICAL TRIAL: NCT04581096
Title: Evaluation of the Response of COVID-19 Spread With a Spatiotemporal Analysis in a Tertiary Hospital
Brief Title: Mapping COVID-19 Spread in a Tertiary Hospital
Acronym: MEDyMAP
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario de Valencia (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Carolina Soledad Romero Garcia, MD, PhD, Anesthesia and Critical care consultant, Hospital General Universitario de Valencia
Other Study IDs: COVID19-MAPA
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Covid19; Spatial Visualization; Neural Network; Respiratory Disease; Pandemic; Disease Spread
MeSH Terms: conditions — COVID-19; Spatial Navigation; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — just descriptive analysis of clinical data

SUMMARY:
One of the major problems in suppressing the spreading of an epidemic resides in understanding and monitoring its propagation patterns, and in evaluating how these are modified by enforced policies. The standard solution requires detailed information at the microscopic scales, e.g. how infected people have moved and whom they came in contact with, which is hardly ever available. The researchers propose a novel approach to the study of the propagation of COVID-19, in which a proxy of this information is derived at macroscopic scales. This will be based on two ingredients: the spatiotemporal study in shiny with mathematical models with aggregated or non aggregated data and the reconstruction of functional networks of spreading patterns, and the development of a supporting software.

ELIGIBILITY:
Inclusion Criteria:

* positive test (PCR or serology) for SARS-CoV-2
* outpatient follow-up

Exclusion Criteria:

* hospitalisation in ward or ICU

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a positive test (PCR or serology) for SARS-CoV-2 in an outpatient regime system
Sampling Method: Non-Probability Sample
Enrollment: 2646 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
spatiotemporal spread | February 1, 2020 to September 30, 2020
  spatiotemporal spread of COVID-19 patient in our hospital

SECONDARY OUTCOMES:
classification score | February 1, 2020 to September 30, 2020
  risk classification score of each patients with clinical and analytical variables

CONTACTS AND LOCATIONS:
Locations (1):
- CHGUV, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
there is not ipd sharing planned

REFERENCES:
- [Background] Romero Garcia C, Iftimi A, Briz-Redon A, Zanin M, Otero M, Ballester M, de Andres J, Landoni G, de Las Marinas D, Catala Bauset JC, Mandingorra J, Conca J, Correcher J, Ferrer C, Lozano M. Trends in Incidence and Transmission Patterns of COVID-19 in Valencia, Spain. JAMA Netw Open. 2021 Jun 1;4(6):e2113818. doi: 10.1001/jamanetworkopen.2021.13818. PMID 34143191
- [Background] Briz-Redon A, Iftimi A, Correcher JF, De Andres J, Lozano M, Romero-Garcia C. A comparison of multiple neighborhood matrix specifications for spatio-temporal model fitting: a case study on COVID-19 data. Stoch Environ Res Risk Assess. 2022;36(1):271-282. doi: 10.1007/s00477-021-02077-y. Epub 2021 Aug 18. PMID 34421343